CLINICAL TRIAL: NCT05174559
Title: Can Care of Adult PKU Be Improved With Additional Dietary Large Neutral Amino Acids: An N-of-1 Study
Brief Title: Additional Dietary Large Neutral Amino Acids (LNAA) for Improved Symptoms in Adult Classical Phenylktonuria (PKU)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: National PKU Alliance (Unknown)
Responsible Party: Principal Investigator, Shoji Yano, Director, Genetics Division, Department of Pediatrics, Associate Professor of Clinical Pediatrics and Medicine, Keck School of Medicine, LAC+USC Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LNAA for PKU
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Phenylketonurias
Keywords: N-of-1 randomized controlled trials
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials in individual patients (interventional N-of-1 RCTs) offer an alternative research design to parallel group randomized controlled trials. The N-of-1 study attempts to determine the more effective treatment for one patient using multiple crossovers, with repetition providing statistical power.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active LNAA (Active Comparator): Active LNAA tablets are given to each participant in 3 multiple crossovers for a total exposure to the Active Comparator 3 times. The allocation is randomized within each cycle of two treatments (active/inactive). There are 3 total cycles for each participant. The intervention is PreKUnil® tablets.
  Interventions: Other: PreKUnil® LNAA Medical Food for PKU
- Inactive LNAA (Placebo Comparator): Inactive LNAA tablets (placebos) are given to each participant in 3 multiple crossovers for a total exposure to the Inactive Comparator 3 times. The allocation is randomized within each cycle of two treatments (inactive/active). There are 3 total cycles for each participant. The placebo intervention is PreKUnil® placebo tablets.
  Interventions: Other: PreKUnil® LNAA Medical Food for PKU

INTERVENTIONS:
Other: PreKUnil® LNAA Medical Food for PKU — PreKUnil® LNAA Medical Food for PKU is a commercially available active LNAA treatment product for PKU. PreKUnil® inactive LNAA is a customized placebo for this research.

SUMMARY:
This research investigates the effects of combining a phenylalanine restricted diet (usual care) with LNAA supplementation (adjuvant LNAA) in well-controlled adults with classical PKU. The hypothesis is that symptoms are improved in well-controlled patients who receive adjuvant LNAA therapy compared with diet monotherapy. Six symptomatic classical PKU adults will be enrolled to test the hypothesis in a small series of N-of-1 randomized controlled trials over 18-weeks. All assessments will be collected in patient's homes. A 3-month follow-up period will assess the longer-term effects of adjuvant LNAA in patients who show clinical benefit at the end of the intervention period.

DETAILED DESCRIPTION:
Clinical care of PKU confronts an increasing proportion of early-treated well-controlled adults, with a treatment goal that quality of life be as normal as possible. Even adults who have successfully managed their blood phenylalanine levels from birth can have symptoms which impact daily function. New therapies that target symptoms are needed, especially for symptomatic well-controlled classical adults with few treatment options. In Denmark and the LAC+USC U.S. clinic, adults are offered large neutral amino acid (LNAA) supplements when diet monotherapy becomes less effective for symptom management, or the patient wants a less restrictive diet. Many patients report improved symptoms. LNAA supplementation doesn't significantly reduce blood phenylalanine, suggesting a different mechanism for patient perceived benefits. Both LNAA supplementation and a phenylalanine restricted diet aim to improve brain neurotransmitter biochemistry to optimize outcomes through dietary intervention. The overall objective of this research is to evaluate additional dietary LNAAs on symptom management in adults with classical PKU at an individual level. N-of-1 randomized controlled trials will provide the highest level of evidence. The scientific premise is that manipulation of dietary LNAAs affects blood LNAA concentrations. LNAAs compete with phenylalanine for a shared transporter from blood to brain, dependent on blood concentrations and transporter affinities. Higher blood phenylalanine levels in adult PKU, with high transport affinity, produces excessive phenylalanine brain entry at the expense of other LNAAs. Insufficient LNAAs impairs synthesis of chemicals in the brain (neurotransmitters), a suggested mechanism of action for adult PKU symptoms. Additional dietary LNAAs may help to overcome this limitation of adult usual care. The study uses established PKU treatment products (medical foods) and biomarkers, (1) to determine effect of the adjuvant LNAA diet in symptom management; and (2) to evaluate correlations between changes in biomarkers and changes in symptoms during the intervention. Should findings show additive clinical value of LNAAs to the PKU diet, the strategy may become a useful adjunct. For participants, results will bring them closer to evidence-based individualized care. This work could advance the field closer toward personalized management.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of classical PKU (blood phenylalanine ≥1200 µmol pre-treatment or off-treatment
* ≥ 2 PKU-related symptoms with clinically meaningful negative impact on daily life
* is in regular clinical monitoring and is treated with a PKU diet with a natural protein restriction and medical foods
* average blood phenylalanine levels between 360 and 900 µmol in past one year
* able and willing to provide consent
* demonstrates capacity to complete all requirements of the protocol
* if on medications approved by the Principal Investigator agrees not to alter dose for duration of study
* has stable daily access to phone, internet, and physical address

Exclusion Criteria:

* women who are breastfeeding, pregnant or planning to become pregnant in the next year
* use of adjuvant PKU treatments (LNAAs, Kuvan®, Palinziq®) within past 3 months
* use of psychotropic medications, melatonin, or any serotonin-reuptake inhibitors within past 3 months
* demonstrates insufficient motivation or time required to complete full trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Personalized Symptom Index | 3 weeks
  Assesses the subjective effect of the interventions on the personally relevant two most bothersome symptoms for the individual patient as identified in a Symptom Elicitation Interview

SECONDARY OUTCOMES:
Absolute plasma phenylalanine concentration, dried blood spots (finger-prick method) | 3 weeks
  Primary FDA-qualified biomarker for PKU
Fasting plasma LNAAs, dried blood spots (finger-prick method) | 3 weeks
  Secondary biomarkers such as the plasma Phe/Tyr ratio, Tyr/LNAA, Trp/LNAA ratio
Urine peripheral biomarkers of neurotransmitters, dried urine spots | 3 weeks
  6-sufatoxymelatonin and dopamine
Computerized neuropsychological testing (responses over study iPad from home) | 3 weeks
  Cambridge Neuropsychological Test Automated Assessment Battery (CANTAB) customized for study
PKU-QOL Questionnaire Adult version (responses over study iPad from home) | 3 weeks
  65-item (20 min) Patient-Reported Outcome Measure of the impact of PKU and the PKU diet on quality of life
Psychological General Well-Being Index (responses over study iPad from home) | 3 weeks
  22-item (15 min) Patient-Reported Outcome Measure of well-being
Adult ADHD Self-Report Scale (ASRS v1.1) | 3 weeks
  9-item inattention subscale (10 min) Patient-Reported Outcome Measure of attention
3-Day Diet Record | 3 weeks
  Complete recording of 24-hr intake for 3 days (45 min)

CONTACTS AND LOCATIONS:
Overall Officials: Shoji Yano, MD, PhD, Principal Investigator — Keck School of Medicine at USC
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No